CLINICAL TRIAL: NCT06751836
Title: Advancing Pandemic Preparedness: Innovative Multidisciplinary Strategies for COMBATing Severe Dengue
Brief Title: Innovative Multidisciplinary Strategies for Combating Severe Dengue
Acronym: COMBAT
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: BIO BOX GUATEMALA ONG DE INVESTIGACIÓN, SERVICIOS Y DE MEDIO AMBIENTE (Unknown); DEVKI DEVI FOUNDATION SOCIETY, India (Unknown); MANIPAL ACADEMY OF HIGHER EDUCATION, India (Unknown); Artemis Medicare Services Ltd., India (Unknown)
Responsible Party: Principal Investigator, Ujjwal Neogi, Senior Lecturer, Karolinska Institutet
Other Study IDs: COMBAT (2024-05758-01); 101191315 (Other Grant/Funding Number: European Commission:European Health and Digital Executive Agency (HADEA))
Record Dates: First submitted 2024-12-13; First posted 2024-12-30 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-12

CONDITIONS: DENV Without Warning Signs; DENV with Warning Signs; Severe Dengue; Healthy Controls Group - Age and Sex-matched
Keywords: Severe Dengue; Multi-omics; Predictive biomarker
MeSH Terms: conditions — Severe Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Dengue without warning signs (DwoWS): Laboratory confirmed Dengue without plasma leakage
  Interventions: Other: Infection and no infection
- Dengue with warning signs (DWS): Laboratory confirmed Dengue without plasma leakage plus abdominal pain, persistent vomiting, fluid accumulation, mucosal bleeding, lethargy, liver enlargement, increasing haematocrit with decreasing platelets
  Interventions: Other: Infection and no infection
- Severe Dengue (SD): Dengue with severe plasma leakage, severe bleeding, or organ failure
  Interventions: Other: Infection and no infection
- Healthy Control: Healthy participants who have tested negative for dengue infection

INTERVENTIONS:
Other: Infection and no infection — No intervention apart from the dengue infection
  Groups: Dengue with warning signs (DWS); Dengue without warning signs (DwoWS); Severe Dengue (SD)

SUMMARY:
The goal of this observational study is to identify biomarkers and host factors associated with dengue severity in patients from dengue-endemic regions. The main question it aims to answer is:

Can multi-omics approaches predict disease severity and identify key factors contributing to severe dengue infections?

Participants will include individuals with dengue infection, and the study will analyze their blood samples using multi-omics techniques to uncover host immune responses, disease pathogenesis, and cellular pathway interactions. The study will also assess the role of primary and secondary infections, virus serotypes, and immunological factors in disease progression. Findings aim to support disease management, improve severity prediction, and identify potential therapeutic targets to prevent severe outcomes.

DETAILED DESCRIPTION:
Background: Many ongoing dengue clinical trials aim to evaluate both therapeutic compounds and potential vaccine candidates. The therapeutic compounds aim to target various stages of dengue virus replication, such as viral entry, by inhibiting virus fusion, NS5 polymerase inhibitor, and NS1 antigenemia reduction, to mention a few. However, an omics-based approach to identifying the metabolic pathways that dengue utilizes to subvert the host system to derive energy from and subsequently deploy viral immune evasion strategies has yet to be established. This study will focus on exploring and understanding the pathways that the dengue virus exploits and investigate if blocking the identified pathway can cause the virus to 'starve.'

* The study will offer insight into the diverse system-level range of dengue infection markers and the dysregulated molecules involved in cellular and metabolic pathways during dengue infection.
* The identification of novel pathways affected by molecule dysregulation will unveil the association of the biomarkers with immune response and disease severity, thereby helping to improve patient triage and treatment.
* The identified biomarkers will be significant in monitoring patients, creating a platform for early intervention to mitigate severe dengue through novel therapeutic targets and management strategies.

The primary objectives of the proposed study are:

* Case-wise viral serotyping and investigation of host cytokine profile.
* System-wide blood-transcriptomics and proteomics during dengue infection and its relationship with disease severity.
* Identification of pathways influencing severity by in vitro mechanistic studies.

Study Cohorts:

Clinical material from two endemic regions, one from Central America (Guatemala) and Southeast Asia (India) will be used. Guatemala is an exemplary location for studying the DENV infection, owing to its distinctive combination of climatic diversity and endemic and dengue presence. Two blood samples (on the day of hospitalization and the day of discharge) from the patients will be collected as per the WHO revised 2009 case classification: 1) dengue without warning signs (DwoWS, n=200), 2) dengue with warning signs (DWS, n=200), 3) severe dengue (SD, n=200). Additionally, non-dengue samples will be collected from healthy controls (n=200). This cohort will act as the DISCOVERY cohort. We will collect whole blood in a TempusTM tube (for RNA sequencing) and serum (for proteomics and metabolomics).

Under the India-EU cooperation on research & innovation (R&I) and co-funding partnership under the EU framework program on R&I 'Horizon Europe, samples will be collected from India, from Artemis Hospital, New Delhi, Max Health Care, New Delhi (a unit of Devki Devi Foundation) and Kasturba Medical College Hospital, Mangalore. Those are the two epicentres of the dengue endemic in India. 50 samples from each dengue severity classification (total samples 150 in each category) and DENV-negative healthy control (total 150: 50 in each site) will be collected. The Indian cohorts will act as the VALIDATION cohorts.

Recruitment of controls Healthy participants who have tested negative for dengue infection in the past three months will not be recruited to the study, which will be further age-and gender-matched with the cases. These samples will be tested for anti-dengue IgM and NS1 ELISA to rule out ongoing asymptomatic infection. They will also be subjected to anti-dengue IgG ELISA to check for past dengue infection. Each of the control participants will also be asked to provide a detailed medical history

ELIGIBILITY:
Inclusion Criteria:

Group 1: Dengue without warning signs Patients presenting with the following symptoms confirmed positive for dengue infection by lab diagnosis by anti-dengue IgM or NS1 ELISA will be recruited for the study under this cohort.

Symptoms will be fever along with at least two of the following -

* Myalgia, arthralgia
* Nausea and/or vomiting
* Rashes
* Leukopenia Group 2: DENV with warning signs This cohort will include patients with the above symptoms and any of the following clinical signs.
* Abdominal pain with tenderness
* Persistent vomiting
* Fluid accumulation
* Mucosal bleeding
* Restlessness, lethargy
* Liver enlargement >2cm
* Laboratory findings: An increase in hematocrit levels and a rapid decrease in platelet count Group 3: Severe dengue
* Severe plasma leakage leads to hypovolemic shock (dengue shock syndrome) and fluid accumulation with respiratory distress.
* Severe bleeding, such as epistaxis, internal bleeding, etc., is evaluated by a clinician.
* Severe organ involvement with any of the following symptoms
* Liver AST or ALT ≥ 1000
* CNS: impaired consciousness
* Heart and other organs failure

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients who are pregnant, immunocompromised, or undergoing chemotherapy, on steroids or immunosuppressive drugs in the last year, liver cirrhosis, or coinfection with a non-dengue pathogen.
  * Cases with a lab-confirmed dengue infection within the past three months will excluded from the case cohort.
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
DISCOVER predictive biomarkers and AI tool for Dengue Severity | From enrollment to the end of hospitalisation at 2 weeks
  This project aims to identify prognostic plasma protein biomarkers for disease severity in dengue virus (DENV) using data from a clinical cohort in an endemic region experiencing a surge in DENV morbidity and mortality.
  It involves developing a novel consensus association-based gene/protein cooperation network to uncover key host factors driving severe disease. Additionally, the project seeks to create AI-driven prognostic tools for predicting DENV severity by integrating patient demographic and clinical data with gene and protein biomarkers, DENV serotyping, and climate information.

CONTACTS AND LOCATIONS:
Locations (2):
- Bio Box Guatemala Ong de Investigación, Servicios Y de Medio Ambiente, Guatemala City, Guatemala
- Manipal Academy of Higher Education (MAHE), Mangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided
Annonymised and delinked IPD can be shared after the completion of the study after getting approval from the steering board and obtaining the ethical clearance of the requesting party.

REFERENCES:
- [Background] Bhatt P, Varma M, Sood V, Ambikan A, Jayaram A, Babu N, Gupta S, Mukhopadhyay C, Neogi U. Temporal cytokine storm dynamics in dengue infection predicts severity. Virus Res. 2024 Mar;341:199306. doi: 10.1016/j.virusres.2023.199306. Epub 2024 Jan 6. PMID 38176525